CLINICAL TRIAL: NCT05422781
Title: A Phase I, Open Label, First In Humans (FIH), Study To Evaluate The Safety, Tolerability And Immunogenicity Of 4 mg Of ITI-3000 In Patients With Polyomavirus-Positive Merkel Cell Carcinoma (MCC)
Brief Title: Study To Evaluate The Safety, Tolerability And Immunogenicity Of 4 mg Of ITI-3000 In Patients With Polyomavirus-Positive Merkel Cell Carcinoma (MCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunomic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITI-3000
Record Dates: First submitted 2022-06-01; First posted 2022-06-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants With Polyomavirus-Positive Merkel Cell Carcinoma (MCC) (Experimental): Eight participants with MCC (> 1.0 years since definitive treatment or participants who had recurrence >2 years since evidence of disease) and NEAD
  Interventions: Drug: ITI-3000

INTERVENTIONS:
Drug: ITI-3000 — ITI-3000 is a DNA vaccine (L-H LT S220A) which contains sequences for both LAMP1 and LTS220A, the truncated form of the LT antigen of MCPyV with a detoxifying serine to alanine mutation at position 220

SUMMARY:
This Phase I clinical trial will evaluate the safety, tolerability, and immunogenicity of 4 mg doses of ITI-3000 in participants with polyomavirus-positive Merkel cell carcinoma (MCC).

DETAILED DESCRIPTION:
This is a single dose design examining 4 mg dose of the DNA vaccine ITI-3000 in participants who were diagnosed with polyomavirus-positive MCC, histologically confirmed by an expert pathologist on standard clinical staining, that may have been supplemented by specific staining for Cytokeratin 20 (CK20) and/or other markers used to distinguish MCC.

Evidence of Merkel cell polyomavirus (MCPyV) in the tumor at initial presentation (pre-therapy) can be provided by a positive anti-MCPyV oncoprotein antibody AMERK Test.

Participants in the study are those who are both diagnosed and have completed standard of care (SOC) surgical and/or radiation therapy at least 1 year prior to enrollment in the study and have no evidence of active disease (NEAD). Participants those who were previously diagnosed with MCC, and had recurrence and also exhibited no evidence of active disease (NEAD) for more than 2 years prior to enrollment in the study.

NEAD is confirmed by physical examination, a negative AMERK test (<74 STU) in participants with a prior positive AMERK test, or significantly decreased, stable AMERK titers in 2 or more consecutive draws compared to prior positive AMERK test at the time of diagnosis, in the setting of a negative computed tomography (CT) scan of the chest, abdomen and pelvis or PET-CT within 3 months of enrollment into the study.

Eight participants will be enrolled at 4 mg total DNA dose to assess safety, tolerability, and immunologic response to the ITI-3000 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Merkel cell polyomavirus (MCPyV) in the tumor at initial presentation (pre-therapy) can be provided by a positive anti-MCPyV oncoprotein antibody AMERK Test.
* Eligible participants have to be both be diagnosed and have completed SOC surgical and/or radiation therapy at least 1 year prior to enrollment in the study and have no evidence of active disease (NEAD).
* Participants who were previously diagnosed with MCC and had recurrence and also exhibited no evidence of active disease (NEAD) for more than 2 years prior to enrollment in the study.
* Age ≥ 18 years.
* Karnofsky performance status (PS) ≥ 70 or ECOG PS 0-1.
* Participant has a predicted life expectancy ≥ 3 months.
* Participant provided signed and dated informed consent prior to initiation of any study procedures.
* Participant has adequate renal function (creatinine ≤ 1.5 times the upper limit of normal [ULN]) or a glomerular filtration rate (GFR) of ≥ 50 mL/min/1.73 m2).
* Participant has adequate hepatic function, as evidenced by a total bilirubin ≤ 1.5 times the ULN, aspartate transaminase (AST), and/or alanine transaminase (ALT) ≤ 3 times the ULN.
* Participant has adequate bone marrow function, as evidenced by hemoglobin ≥ 9.0 g/dL in the absence of transfusion within the previous 72 hours, platelet count ≥ 100×109cells/L, and absolute neutrophil count (ANC) ≥ 1.5×109 cells/L.
* Participant and his/her partner agree to use adequate contraception after providing written informed consent through 2 months after the last study drug dose, as follows:

  * For women: Negative pregnancy test during Screening and at Baseline and compliant with two methods of medically-approved contraceptive regimens or abstinence during and for 2 months after the treatment period or documented to be surgically sterile or postmenopausal.
  * For men: Compliant with two methods of medically approved contraceptive regimens or abstinence during and for 2 months after the treatment period or documented to be surgically sterile
* Participant is willing and able to participate in the study and comply with all study requirements.

Exclusion Criteria:

* Participation in another therapeutic clinical trial.
* Participant who received systemic treatment previously (e.g., chemotherapy, PD-1/PD-L1).
* Participant is pregnant or breast-feeding.
* Negative for an anti-MCPyV oncogene antibody titer or other evidence of no MCPyV involvement at initial presentation using an acceptable and specific assay at the institution.
* Known history of AIDS/HIV, other viral diseases or oncologic disorders such as untreated HCV, chronic active HBV or organ transplantation that may have immunologic consequences or require immunosuppression. No testing required.
* Participant with CLL-associated MCC.
* On-going immunosuppressive therapy for other conditions with the exception of low-dose topical, nasal or inhaled steroids.
* Participant has a history of other malignancy treated with curative intent within the previous 3 years with the exception of adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix. Participants with previous invasive cancers are eligible if the treatment was completed more than 3 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
* Participant has a significant medical illness or abnormal laboratory finding that, in the Investigator's opinion, would increase the risk of participating in this study.
* Participant with otherwise unexplained >10% weight loss in the last 30 days prior to the screening.
* Participant has evidence of serious active infection (i.e., infection requiring treatment with intravenous antibiotics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs). | Through study completion, up to 12 months.
  Number of participants that experience any Dose Limiting Toxicities (DLTs).
Number of occurrences of Adverse events/Serious Adverse Events that will be assessed for severity according to the NCI CTCAE, version 5.0. | Through study completion, up to 12 months.
  Number of occurrences of Adverse events/Serious Adverse Events that will be assessed for severity according to the NCI CTCAE, version 5.0.
Number of participants with changes from baseline in physical exam findings. | Through study completion, up to 12 months.
  Number of participants with changes from baseline in physical exam (e.g. weight, height, etc.) findings.
Number of participants with changes from baseline in hematology lab results. | Through study completion, up to 12 months.
  Number of participants with changes from baseline in hematology lab results (e.g. Hgb, PLT CT, Hct, RBC, etc.).
Number of participants with changes from baseline in chemistry lab results. | Through study completion, up to 12 months.
  Number of participants with changes from baseline in chemistry lab results (e.g. Alb, ALK, CO2, BUN, Glu,etc.) .
Number of participants with changes from baseline in urinalysis lab results. | Through study completion, up to 12 months.
  Number of participants with changes from baseline in urinalysis lab results (e.g. SPG, pH, TP, Glu, etc.) .
Number of participants with changes from baseline vital signs. | Through study completion, up to 12 months.
  Number of participants with changes from baseline vital signs (e.g. body temp, BP, RR, etc.) .

OTHER OUTCOMES:
Exploratory endpoints include immune assessments for anti-MCPyV T-cell response | Through study completion, up to 12 months.
  Changes in titers from baseline.
Exploratory endpoints include immune assessments anti- MCPyV LT antibodies | Through study completion, up to 12 months.
  Changes in titers from baseline.
Exploratory endpoints include immune assessments for anti-MCPyV oncoprotein antibodies | Through study completion, up to 12 months.
  Changes of anti-MCPyV oncoprotein antibodies from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington/Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchta Rosean C, Leyder EC, Hamilton J, Carter JJ, Galloway DA, Koelle DM, Nghiem P, Heiland T. LAMP1 targeting of the large T antigen of Merkel cell polyomavirus results in potent CD4 T cell responses and tumor inhibition. Front Immunol. 2023 Aug 30;14:1253568. doi: 10.3389/fimmu.2023.1253568. eCollection 2023. PMID 37711623